CLINICAL TRIAL: NCT06510439
Title: Randomized, Controlled Trial of Need to be Needed (N2BN) Intervention to Improve Social Connection, Reduce Social Isolation and Loneliness
Brief Title: Need to be Needed (N2BN) Intervention
Acronym: N2BN RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 90DPCp0011-01-00; 31409 (Other: Temple University)
Record Dates: First submitted 2024-07-14; First posted 2024-07-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Loneliness; Social Isolation
Keywords: mattering; loneliness; social isolation; need to be needed; neededness; volunteering
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and research assistant completing baseline, mid-point and end-point interview are blind to treatment allocation. Data analyst will be blind to participant condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Need to be Needed Intervention (Experimental): Interventionists will meet with participants to discuss supported volunteering concepts and develop an initial plan. This plan will be flexible as it is likely that participants will need multiple opportunities to identify and explore options for voluntarism. Once the plan is developed, interventionist will make weekly contact to support participants in achieving goals. These weekly contacts (3x per month) are expected to be brief (30-40 minutes) and focused on information sharing and supported problem solving. Interventionists will also schedule monthly plan reviews (1x per month) with participants to review and revise supported volunteering individualized plans. Both clients who are achieving goals as well as those falling short of their goals may want to revise or change their plan.
  Interventions: Behavioral: Need to Be Needed Intervention
- Active control group (Active Comparator): Participants assigned to the attention control condition will receive printed information on the importance and opportunities for volunteering and will be encouraged to review resources from the TU Collaborative website. They will receive weekly 10-minute non-directive supportive listening sessions via telephone/videoconferencing with a Research assistant. Research assistants are full-time staff members with an undergraduate degree in psychology. Undergraduate students are not involved in performing the weekly check-ins with the control group. The control group will not receive weekly 1:1 support through a trained clinician.
  Interventions: Other: Active Control Group

INTERVENTIONS:
Behavioral: Need to Be Needed Intervention — Interventionist-supported volunteering intervention that targets opportunities creating social connections that matter through focus on kindness and gratitude throughout the intervention.
  Other Names: N2BN Intervention
  Arms: Need to be Needed Intervention
Other: Active Control Group — Weekly non-directive listening support
  Arms: Active control group

SUMMARY:
The proposed study is a randomized, controlled trial (RCT) that will examine the effectiveness of an intervention designed to reduce social isolation and loneliness of adults with serious mental illness (SMI). The intervention will focus on improving their sense of mattering by using acts of kindness and experiencing gratitude through volunteering. 120 participants will be randomly assigned to the intervention group or the attention control group. Over the course of the 6-month intervention, participants in the intervention arm, will receive weekly support from the interventionist. The interventionist and the participant will collaboratively set goals and develop an initial intervention plan, which is informed by the participants interests, values and goals. The attention control group will receive non-directive listening support through research assistants.

Data collection for all participants will occur at baseline, at the mid-point of the intervention at 3 months, and at the end of the 6-month intervention. Participants will be asked questions about quality of experience, social context and satisfaction, mattering components, kindness, gratitude, and loneliness. We will gather data on demographic background, life transitions, social network characteristics, internalized stigma, neighborhood climate, depression, and trait measures of mattering and loneliness during intake and exit interviews. Additionally, participants of the intervention arm will be asked to provide feedback about the intervention.

DETAILED DESCRIPTION:
The proposed study is a randomized, controlled trial (RCT) that will examine the effectiveness of an intervention designed to reduce social isolation and loneliness of adults with serious mental illness (SMI) receiving community mental health services. Specifically, the intervention will focus on improving their sense of mattering by using acts of kindness, and experiencing gratitude through volunteering.

This intervention is based on evidence-based models and takes a different approach than many loneliness and social connectedness interventions. Using the CIVIC Framework and Mattering Wheel as a foundation, this intervention has the potential to develop relationships of equality and reciprocity that extend beyond the intervention period. This intervention also draws upon our own intervention research which utilized the Individualized Placement and Support model in a supported leisure intervention.

Participants will be randomly assigned to the intervention group or the attention control group. Those in the intervention arm receive weekly support of an interventionist leading the intervention which is based on the aforementioned frameworks and informed by the idiosyncratic experiences and values of the participant. The control group will receive weekly non-directive listening support through research assistants and printed information on the importance, skills, and opportunities for participation.

Over the course of the 6-month intervention, participants in the intervention arm, will receive weekly support from the interventionist. The interventionist and the participant will collaboratively set goals and develop an initial intervention plan, which is informed by the participants interests, values and goals. Participants will receive support through weekly meetings through the interventionist who will monitor their progress, assist with problem solving and facilitates changes as needed. The attention control group will receive weekly non-directive listening support through research assistants.

Recruitment will occur only in Philadelphia in collaboration with outpatient treatment service providers. Data collection for all participants will take occur at baseline, at the mid-point of the intervention at 3 months, and at the end of the 6-month intervention.

The overall objective of the current study is to evaluate the outcomes associated with the Need to be Needed intervention. This project aims to address the following research questions:

RQ1a. Is participation in the intervention associated with reductions in loneliness? RQ1b. Is participation in the intervention associated with reductions in social isolation? RQ2. Are improvements in intervention targets (mattering, kindness, gratitude) predictive of social isolation and loneliness outcomes? RQ3. Is the intervention acceptable to individuals with SMI? RQ4. Is the implementation of this intervention feasible?

Group Assignment

Once participants have completed the informed consent process and baseline data collection, they will immediately be randomly assigned either the intervention or control group. Randomization will be done in blocks of ten by assigned participant number (i.e., #1 to #120) to prevent runs and enhance the probability of creating comparable groups.

N2BN Intervention

The proposed Need to be Needed (N2BN) intervention is a 6-month, supported volunteering intervention that targets opportunities creating social connections that matter through focus on kindness and gratitude throughout the intervention. At the beginning of the intervention, the interventionist will work with the participant to explore interests and identify opportunities for volunteering. The exploration of interests and interest-based opportunities supports the participants' autonomy and maximizes the benefits of volunteering. Part of this exploration includes the identification of welcoming places using the tools developed by the Temple University Collaborative on Community Inclusion. Welcoming places will then be explored to determine whether there are opportunities for volunteering within those locations. Encouraging participants to volunteer in places where they already feel welcome may more rapidly facilitate engagement in volunteering and enhanced social connectedness.

The chosen volunteer location must provide opportunity for consistent and sustained participation. Participants will be encouraged and assisted by interventionist to identify a volunteer opportunity that would allow for at least weekly engagement. Once a location is identified, the interventionist will work with the participant to identify the necessary skills for volunteering in that role. Consistent with the IPS model, these skills will be practiced and refined while volunteering at the chosen site. Each week, the interventionist will meet with the participant to discuss the activities done while volunteering and how those activities contributed to the overall success of the program. Additionally, the interventionist will facilitate discussions about the people at the volunteer site and explore opportunities for relationship development.

Because kindness and gratitude contribute to increases in social connectedness, we will include opportunities to engage in and document acts of kindness and feelings of gratitude. Throughout the first half of the intervention, the participant will be encouraged to identify acts of kindness he or she engages in at the volunteer location. This could include the volunteer activity alone or may include random acts of kindness that the participant initiates (e.g., helping beyond the volunteer time, offering to help another volunteer with something, bringing someone a coffee 'just because,' among others).

Participants will then be encouraged to expand these acts of kindness to their broader community. This will start with opportunities to engage in random acts of kindness within ones' welcoming places and then move to other community locations and relationships. Participants will be encouraged to practice kindness within the four areas (I.e., community, commitments, relationships, and self) of the mattering wheel. This provides an opportunity for participants to 'add value' to multiple life domains.

In the last half of the intervention, participants will be introduced to the concept of gratitude and engaging in intentional expressions of gratitude. Many interventions use writing as a strategy to document and express gratitude. This includes letter writing, journaling, and writing social media posts. Similarly, this intervention will encourage participants to create a gratitude journal and also encourage participants to express their gratitude to others- via writing or other means of communication. Participants will be encouraged to focus their journaling on gratitude related to individuals with whom they have either developed relationships or interacted with during the course of the intervention. Similarly, participants will be encouraged to document and express gratitude within the four areas (I.e., community, commitments, relationships, and self) of the mattering wheel. This process allows participants to explore and document the 'value gained.' Additionally, the participant and interventionist will discuss how the feelings of gratitude may lead to additional acts of kindness or ways to give back to the relationship.

Throughout the intervention, the interventionist will work closely with the participant to develop an individualized supports plan. This may include developing a visual calendar to support engagement in the volunteer activities; identifying natural supports to encourage ongoing participation; or scheduling opportunities for touring the volunteer location prior to volunteering, among others. Many of these strategies were developed and used by our team when implementing a supported leisure intervention. Additionally, the interventionist will talk with the participant weekly about potential social connections and navigate strategies to nurture those potential relationships.

Intervention frequency, intensity and duration. Interventionists will meet with participants initially to discuss supported volunteering concepts and develop an initial plan. It is anticipated that this initial contact will require 2-3 hours of time and may occur in more than a single meeting. This plan will be flexible as it is likely that participants will need multiple opportunities to identify and explore options for voluntarism. Once the initial plan is developed, the interventionist will make weekly contact either in person or via telephone/videoconference to support participants in achieving goals. These weekly contacts (3x per month) are expected to be brief (30-40 minutes) and focused on information sharing and supported problem solving. Interventionists will also schedule monthly plan reviews (1x per month) with participants to review and revise supported volunteering individualized plans. Both clients who are achieving goals as well as those falling short of their goals may want to revise or change their plan. Over the course of the 6-month intervention, it is projected that interventionists will engage with participants numerous times, possibly up to 40-45 hours of contact. Based on the planned enrollment of 10 participants per month, with five randomized into the treatment condition, the maximum number of individuals who could be supported per FTE navigator would be 20 participants. This consumer/staff ratio is below what is typically seen in such services as supported employment or education.

Control group

Participants assigned to the attention control condition will receive printed information on the importance and opportunities for volunteering and will be encouraged to review resources from the TU Collaborative website. They will receive weekly 10-minute non-directive supportive listening sessions via telephone/videoconferencing with a Research assistant. Research assistants are full-time staff members with an undergraduate degree in psychology. Undergraduate students are not involved in performing the weekly check-ins with the control group. The control group will not receive weekly 1:1 support through a trained clinician.

ELIGIBILITY:
Inclusion Criteria:

1. A research diagnosis of Major Depression, Bipolar I, II, or Schizophrenia Spectrum disorder.

   Participants will be screened by research staff using sections of the Mini-International Neuropsychiatric Interview (MINI; Sheehan et al., 1998) that will identify research diagnoses of: Major Depression, Bipolar I, II, or Schizophrenia Spectrum disorder.
2. Ages 18 years old and older
3. Living in the community
4. Able to communicate in written and oral English
5. UCLA-Loneliness Scale score of 6 or higher

Exclusion Criteria:

1. Having a legal guardian
2. Unable to give informed consent.
3. Living situation which restricts their ability to move freely

Potential participants failing to meet screening criteria will be informed at the time that we are not able to enroll them in the study at this time. Any interview notes, or information recorded on the MINI will be destroyed or securely deleted.

The study will not enroll any vulnerable populations.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2035-05-31 (Estimated)

PRIMARY OUTCOMES:
Change of Demographic Background | baseline, after 3-months, after 6-months
  Standard personal characteristics will be assessed via intake interview. Demographic items will include 11 items identifying employment, income, marital status
Change of Neighborhood Social Climate Scale from Housing Environment Survey | baseline, after 3-months, after 6-months
  Neighborhood Social Climate Scale from Housing Environment Survey (HES) (Kloos & Shah, 2009): This 12-item subscale from the HES includes questions related to housing type (independent, familial, group), social context (alone, partnered, with others), stability (the length lived at their current residence), and satisfaction with one's housing and neighborhood
Change of Social Network | baseline, after 3-months, after 6-months
  Social Network Generator (Pescosolido & Wright, 2004): This instrument identifies important people connected with the respondent. Network size, composition, contact, closeness, reciprocity, changes will be quantified.
Change of sense of mattering | baseline, after 3-months, after 6-months
  Interpersonal Mattering Scale (Moschella & Baynard, 2021; Elliott et al., 2004): This 12-item scale examines three dimensions of mattering, including awareness (a=.87), importance (a=.89), and reliance (a=86).
Change of sense of loneliness | baseline, after 3 months, after 6 months
  3-Item UCLA Loneliness Scale (Hughes, Waite, Hawkley, & Cacioppo, 2004). This brief measure of loneliness has shown satisfactory reliability and validity in the measurement of overall loneliness. (this instrument is repeated from intake interview)
Change of sense of loneliness | baseline, after 3 months, after 6 months
  6-item DeJong Gierveld Loneliness Scale (De Jong Gierveld & van Tilburg, 2006) This 6-item measure is used to create a unidimensional overall loneliness measure as well as provide information about the emotional and/or social loneliness situation of respondents. Social loneliness reflects dissatisfaction with social relationships, whereas emotional loneliness represents dissatisfaction with a close discussion partner. (this instrument is repeated from intake interview)
Change of depressive symptoms | baseline, after 3 months, after 6 months
  Center for Epidemiological Studies Depression Scale (CES-D; Radloff, 1977): This is a 20-item scale of depressive symptoms covering the prior week. a= .85-.90
Change of sense of emptiness | baseline, after 3 months, after 6 months
  The Psychological Emptiness Scale (PES) Herron et al., (2024) This instrument is a 19-item scale to measure the subjective experience of the sense of emptiness over the past month.
Change of community participation | Baseline, after 3 months, after 6 months
  Temple University Community Participation Measure (TUCP). This measure records self-reports of community participation in 26 different areas including going to a supermarket, participating in a community social group (like a book club or recreational sports team), going to a movie, or working for pay. Participants are asked to indicate the number of days in the past 30 days that they participated in each of the 26 areas, whether each participation area was important to them, and whether they felt they participated in each area enough, not enough, or too much. Recent research has found the measure to be reliable and valid.
Change of health outcome | Baseline, after 3 months, after 6 months
  PROMIS® Scale v1.2 - Global Health- Patient Reported Outcome Measurement Information System (PROMIS) Global Health v1.2 short form is a 10-item instrument representing multiple domains. Scores are assigned for both Global Physical Health component and Global Mental Health component.
Change of perceived stigma | Baseline, after 3 months, after 6 months
  Internalized Stigma of Mental Illness scale (ISMI-10) (Hammer & Toland, 2017): Internalized stigma will be assessed via this 10-item measure that has demonstrated adequate internal consistency, reliability and external validity. The ISMI-10 was found to have a good internal consistency reliability of 0.75.
Change of perceived acts of kindess | Baseline, after 3 months, after 6 months
  Kindness Measure (Young, et al., 2021): Created as a 20-item measure to assess the amount and variety of kindness a person exhibits. Contains subscales of a) affective-socially prescribed, b) anthropophobia, c) affective-proactive, d) principle-socially prescribed, and e) principle-proactive (subscale internal consistency .68-.95).
Change of perceived gratitude | Baseline, after 3 months, after 6 months
  Gratitude Questionnaire (GQ-6) (McCullough et al., 2002)- The Gratitude Questionnaire-Six-Item Form (GQ-6) is a six-item self-report questionnaire designed to assess individual differences in dispositional gratitude in daily life. Respondents endorse each item on a 7-point Likert-type scale (where 1 = strongly disagree and 7 = strongly agree), with two items negatively worded. It demonstrates good internal reliability with alphas between .82 and .87.
Change of overall well being | Baseline, after 3 months, after 6 months
  Overall Well Being PERMA Profile (Butler & Kern, 2016) This instrument is a brief 23-item measure of overall well-being and examines positive emotion, engagement, relationships, meaning and accomplishment, as well as negative emotion and perceived health. The instrument has demonstrated good psychometric properties in large-scale studies with adults. This measure will support identification of important relationships; however, additional domains can be examined in relation to engagement and purpose in life.
Change of recovery assessment | Baseline, after 3 months, after 6 months
  Recovery Assessment Scale (RAS-20): assesses self-determination and hope as it relates to recovery. It is frequently used as an outcome measure for program evaluations. It is a 20-item self-report measure. Items are scored on a 5-point Likert scale and range from strongly agree to strongly disagree
Change of social support | Baseline, after 3 months, after 6 months
  The MOS Social Support survey: a 19-item measure with 4 support scales (Emotional/Informational, Tangible, Affectionate, and Positive Social Interaction) and an overall functional social support index that has been shown to have good reliability and validity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hall Mercer, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All participants in the study will be required to complete informed consent forms which will include a clause about data preservation and sharing. Subjects will be assured that their identity will be protected and that no personally identifiable information (PII) will be disclosed as part of any data sharing.
  All data will be stored on Temple University's password protected, HIPAA-approved secure data server. However, because not all investigators who will need access to the data are at Temple, deidentified, anonymized data may be shared with other investigators via a secure file transfer system.
  All data in the study transferred between Temple University and collaborating institutions will be transferred through TUSafeSend using data encryption by way of a secure socket transfer protocol. TUSafeSend provides a secure method for transferring files containing confidential or other sensitive information, including HIPAA authorized data with PHI or PII.

REFERENCES:
- [Background] Hare-Duke L, Dening T, Oliveira D, Dewa R, Slade M. Social connectedness in adults with mental disorders: ecological validation of a conceptual framework for novel complex interventions. J Ment Health. 2021 Jun;30(3):333-340. doi: 10.1080/09638237.2021.1875409. Epub 2021 Feb 1. PMID 33522341
- [Background] Prilleltensky I. Mattering at the Intersection of Psychology, Philosophy, and Politics. Am J Community Psychol. 2020 Mar;65(1-2):16-34. doi: 10.1002/ajcp.12368. Epub 2019 Aug 13. PMID 31407358
- [Background] Snethen G, McCormick BP, Van Puymbroeck M. Community involvement, planning and coping skills: pilot outcomes of a recreational-therapy intervention for adults with schizophrenia. Disabil Rehabil. 2012;34(18):1575-84. doi: 10.3109/09638288.2011.650315. Epub 2012 Feb 6. PMID 22303816
- [Background] Kim J, Morgul K. Long-term consequences of youth volunteering: Voluntary versus involuntary service. Soc Sci Res. 2017 Sep;67:160-175. doi: 10.1016/j.ssresearch.2017.05.002. Epub 2017 May 13. PMID 28888284
- [Background] Wong YJ, Owen J, Gabana NT, Brown JW, McInnis S, Toth P, Gilman L. Does gratitude writing improve the mental health of psychotherapy clients? Evidence from a randomized controlled trial. Psychother Res. 2018 Mar;28(2):192-202. doi: 10.1080/10503307.2016.1169332. Epub 2016 May 3. PMID 27139595
- [Background] O'Connell BH, O'Shea D, Gallagher S. Feeling Thanks and Saying Thanks: A Randomized Controlled Trial Examining If and How Socially Oriented Gratitude Journals Work. J Clin Psychol. 2017 Oct;73(10):1280-1300. doi: 10.1002/jclp.22469. Epub 2017 Mar 6. PMID 28263399
- See also: N2BN information — https://tucollaborative.org/n2bn/